CLINICAL TRIAL: NCT00945646
Title: A Multi-Center, Randomized, Double-Masked, Vehicle-Controlled Clinical Study Evaluating the Efficacy Of FST-201 (Dexamethasone 0.1%) Otic Suspension in Subjects With Acute Fungal Otitis Externa
Brief Title: FST-201 In The Treatment of Acute Fungal Otitis Externa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FST201-AFOE-02
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Acute Fungal Otitis Externa
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FST-201 (dexamethasone 0.1%) Otic Suspension (Experimental)
  Interventions: Drug: FST-201 (dexamethasone 0.1%) Otic Suspension
- vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: FST-201 (dexamethasone 0.1%) Otic Suspension — Instill four drops times two times a day.
  Arms: FST-201 (dexamethasone 0.1%) Otic Suspension
Drug: Vehicle — Instill four times two times a day
  Arms: vehicle

SUMMARY:
The objective of this study is to evaluate the efficacy of FST-201 compared to vehicle in the treatment of acute fungal otitis externa. This trial is designed to enable filing of a New Drug Application in support of FST-201 for the indication of acute fungal otitis externa.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of AFOE of in one or both ears, based on a clinical score of at least 1 for edema (0-3 scale), 2 for overall inflammation (0-3 scale) and 1 for tenderness (absent=0, present=1) and/or 1 for pruritis (absent = 0, present = 1)
* Have appearance consistent with fungal debris, i.e. white or black appearance consistent with Aspergillus spp. or Candida spp.
* Be at least 18 years of age at Visit 1 (Day 1, Screening/Baseline) of either sex and any race
* Provide written informed consent
* Be willing and able to follow all instructions and attend all study visits
* If female and of child bearing potential, agree to and submit a urine sample for pregnancy testing at Visit 1 and upon their exit from the study. Post menopausal is defined as having no menses for 12 consecutive months.

Exclusion Criteria:

* Have known sensitivity to any component of the study medications
* Have a current infection requiring systemic antimicrobial treatment
* Take any systemic (within 30 days) or otic corticosteroids (within 1 day) prior to Visit 1
* Have used topical or systemic anti-inflammatory agents on the same day as Visit 1 and for the duration of the study
* Have used topical or systemic pain medications on the same day as Visit 1 and for the duration of the study
* Have used any topical otic treatment within 1 days prior to Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

PRIMARY OUTCOMES:
Overall clinical cure as defined by absence of the signs and symptoms of AFOE including ear inflammation, edema, tenderness, pruritis and otic discharge. | 1 year

SECONDARY OUTCOMES:
Microbiological resolution defined as absence of pre-treatment pathogenic fungal species. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - ENT Associates of South Florida, Boynton Beach, Florida
  - Sarasota, Florida
  - Austin Ear, Nose, and Throat Clinic, Austin, Texas
  - San Antonio Ear, Nose, and Throat Research, San Antonio, Texas
  - Ear Institute of Texas, San Antonio, Texas